CLINICAL TRIAL: NCT01154361
Title: A Multicenter Study, Randomized, Double-blind With 2 Groups as Prove of Concept for the Treatment of ACEI Induced Angioedema With Subcutaneous Icatibant
Brief Title: AMelioration of Angiotensin Converting Enzyme Inhibitor Induced Angioedema Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMACE
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Angioedema
Keywords: ACE inhibitor induced angioedema; Bradykinin; Non-itching edema; Non-allergic angioedema; Quincke edema; Drug induced angioedema; Bradykinin B2 receptor antagonist; Icatibant; HOE 140
MeSH Terms: conditions — Angioedema | interventions — icatibant; Injections, Subcutaneous; Cortisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Icatibant (subcutaneous) and plazebo (intravenous)
- Arm B (Active Comparator)
  Interventions: Drug: Cortisone + Clemastin (intravenous) and plazebo (subcutaneous)

INTERVENTIONS:
Drug: Icatibant (subcutaneous) and plazebo (intravenous)
  Arms: Arm A
Drug: Cortisone + Clemastin (intravenous) and plazebo (subcutaneous)
  Arms: Arm B

SUMMARY:
This is a multicenter study recruiting patients with angioedema induced by ACEI.

Open-label treatment with subcutaneous Icatibant compared to a historic group of 47 patients with ACE inhibitor induced angioedema which the investigators have been previously treated in the investigators centers with current "standard" therapy (250 mg methylprednisolon and 2 mg clemastine).

In cases with fast progression of edema after application the study-drug, a second application with icatibant could be necessary. Rescue medication and intervention.

DETAILED DESCRIPTION:
Sudden occurrence of subcutaneous or submucosal non-itchy swelling, so-called angioedema, is a well known side effect of angiotensin-converting enzyme inhibitors (ACEi), which may become life-threatening if the upper airway is involved. To be note, ACEi induced angioedema were always located in the head and neck region.

The pathophysiology of ACE inhibitor (ACEi) induced angioedema most likely resembles that of hereditary angioedema (HAE), i.e. it is mainly mediated by bradykinin induced activation of vascular bradykinin B2 receptors (BKR-2). In contrast to an increased bradykinin generation in HAE, treatment with ACEi decreases the bradykinin degradation in plasma and increases the biological activity of bradykinin.

The current pharmacotherapy of ACEi induced angioedema is not satisfactory. Antihistamines and corticosteroids may be effective in the treatment of urticaria with cutaneous edema and itchy, but are theoretically ineffective and hence superfluous in bradykinin induced angioedema. However, glucocorticoids still belong to the standard treatment of angioedema.

We hypothesized that the BKR-2 antagonist icatibant might be an effective therapy for ACEi-induced angioedema.

Patients with ACEi induced angioedema, located in the upper aero-digestive tract will be randomized and treated either with icatibant and plazebo or cortisone with clemastin and plazebo.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 <85 years
* Patient is currently treated with an ACEI
* Patient must have acute angioedema attack caused by an ACEI
* Treatment should be administrated within 10 hrs after onset by an ACEI
* Patient with angioedema of head and /or neck (face, lips, cheeks, tongue, soft palate/uvula, pharynx and larynx)
* At least one moderate to severe severe angioedema symptom as assessed by the investigator, requiring a medical intervention
* Signed written Informed Consent Form

Exclusion Criteria:

* Diagnosis of angioedema that was not caused by ACEI: e.g. hereditary angioedema (C1-INH deficiency), allergy, anaphylaxis, insect bite, trauma, infection, abscess, tumor, post-radiation or post-operative or processes related to salivary glands and others where it is unlikely that the ACEI is causing the angioedema
* Participation in a clinical trial of another investigational medicinal product (IMP) within 30 days
* Patients with acute urticaria
* Patients with a medical history of any angioedema before taking an ACEI
* Patients with an acute rash or hives in the face or somewhere else
* Unstable angina or acute myocardial infarction
* Acute heart failure
* Serious concomitant illnesses that the physician considers to be a contraindication for participation in the trial
* Pregnancy and/or breast-feeding
* Mental condition rendering the patients, in the opinion of the investigator, unable to understand the nature, scope and possible consequences of the study;
* Unlikely to comply with the protocol, e.g., uncooperative attitude, inability to return for the follow-up visit, or unlikely to complete the study for any reason.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Time to complete resolution of angioedema

CONTACTS AND LOCATIONS:
Overall Officials: Murat Bas, Dr., Principal Investigator — Klinikum rechts der Isar, Hals-Nasen-Ohrenklinik, Ismaninger Str. 22 81675 München
Locations (1):
- Klinikum rechts der Isar Hals-Nasen-Ohrenklinik der TUM, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Bas M, Greve J, Stelter K, Havel M, Strassen U, Rotter N, Veit J, Schossow B, Hapfelmeier A, Kehl V, Kojda G, Hoffmann TK. A randomized trial of icatibant in ACE-inhibitor-induced angioedema. N Engl J Med. 2015 Jan 29;372(5):418-25. doi: 10.1056/NEJMoa1312524. PMID 25629740